CLINICAL TRIAL: NCT05749380
Title: Bioequivalence Study to Evaluate Pharmacokinetics and Safety of AmBisome and DKF-5122 in Indicated Patients and Healthy Adults
Brief Title: Pharmacokinetics and Safety of AmBisome and DKF-5122
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DKF-5122-BE
Record Dates: First submitted 2023-02-16; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Invasive Fungal Infections; Neutropenic Fever
MeSH Terms: conditions — Invasive Fungal Infections; Febrile Neutropenia | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1A(RT) (Other): Patients (AmBisome, DKF-5122)
  Interventions: Drug: AmBisome; Drug: DKF-5122
- 1B(TR) (Other): Patients (DKF-5122, AmBisome)
  Interventions: Drug: AmBisome; Drug: DKF-5122
- 2A(RT) (Other): Healthy subjects (AmBisome, DKF-5122)
  Interventions: Drug: AmBisome; Drug: DKF-5122
- 2B(TR) (Other): Healthy subjects (DKF-5122, AmBisome)
  Interventions: Drug: AmBisome; Drug: DKF-5122

INTERVENTIONS:
Drug: AmBisome — Reference, dose of 3 mg/kg.
Drug: DKF-5122 — Test, dose of 3 mg/kg

SUMMARY:
The purpose of the study is to assess the Safety and Pharmacokinetic Characteristics of AmBisome and DKF-5122

ELIGIBILITY:
Inclusion Criteria:

* Part 1. Patients

  1. Age 19 years and older
  2. Empirical therapy for presumed fungal infection in febrile, neutropenic patients
  3. Voluntarily decided to participate in the study and signed the informed consent form
  4. Having contraception during the study
* Part 2. Healthy subjects

  1. Age 19 to 45 years
  2. Body weight 55 kg or more, within ±20% of the ideal body weight
  3. Having no congenital or chronic disease within the last 5 years.
  4. Voluntarily decided to participate in the study and signed the informed consent form
  5. Having contraception during the study

Exclusion Criteria:

* Part 1. Patients

  1. Clinically significant conditions that may affect the pharmacokinetics of amphotericin
  2. History of diseases that may affect the pharmacokinetics of amphotericin
  3. History of drug abuse
  4. History of hypersensitivity to ingredients of investigational products
  5. Unable to maintain proper contraception
  6. Pregnant or breast-feeding
  7. The following laboratory test results at screening

     * Hemoglobin < 8.0 g/dL
     * Serum Creatinine > 2x the UNL
     * AST or ALT > 10x UNL
     * Systolic blood pressure ≥ 140 mmHg or ≤ 90 mmHg
     * Diastolic blood pressure ≥ 90 mmHg or ≤ 60 mmHg
  8. Before the first administration of investigational products

     * Participation to other clinical trials within 6 months
     * Whole blood donation within 60 days or component within 30 days
     * (Herbal) medicines that may affect the pharmacokinetics of amphotericin within 14 days
     * Grapefruit-containing foods within 7 days
     * Excessive exercise within 7 days
  9. Excessive caffeine and alcohol consumption, or a smoker
  10. Not eligible due to other reasons at the investigator's discretion
* Part 2. Healthy subjects

  1. Clinically significant disorders or a medical history of active cardiovascular, respiratory , kidney, endocrine, hematological, digestive, central nervous system, psychiatric disease, or malignant tumor
  2. Clinically significant conditions that may affect the pharmacokinetics of amphotericin
  3. History of diseases that may affect the pharmacokinetics of amphotericin
  4. History of drug abuse
  5. History of hypersensitivity to ingredients of investigational products
  6. Unable to maintain proper contraception
  7. Pregnant or breast-feeding
  8. The following laboratory test results at screening

     * Hemoglobin < 13.0 g/dL
     * Serum Creatinine > 1.25 x UNL
     * eGFR < 90 mL/min/1.73 m2
     * AST or ALT > 1.25 x UNL
     * Total bilirubin > 1.25 x UNL
     * CPK > 1.5 x UNL
     * Systolic blood pressure ≥140 mmHg or ≤90 mmHg
     * Diastolic blood pressure ≥ 90 mmHg or ≤60 mmHg
     * Arrhythmia
  9. Before the first administration of investigational products

     * Participation to other clinical trials within 6 months
     * Whole blood donation within 60 days or component within 30 days
     * Drugs that induce or inhibit drug metabolism enzymes within 30 days
     * Vaccination within 7 days
     * Prescription drugs, herbal medicines, over-the-counters, or vitamins within 14 days
     * Grapefruit-containing foods within 7 days
     * Excessive exercise within 7 days
  10. Excessive caffeine and alcohol consumption, or a smoker
  11. Not eligible due to other reasons at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 to 93 hr
  Liposome encapsulated amphotericin B of healthy adult
AUClast | 0 to 93 hr
  Liposome encapsulated amphotericin B of healthy adult

SECONDARY OUTCOMES:
Cmax | 0 to 93 hr
  Unbound Amphotericin B of healthy adult
AUClast | 0 to 93 hr
  Unbound Amphotericin B of healthy adult
AUCinf | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of healthy adult
tmax | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of healthy adult
t1/2 | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of healthy adult
CL/F | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of healthy adult
V/F | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of healthy adult
Cmin,ss | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of indication patient
Cav,ss | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of indication patient
tmax,ss | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of indication patient
t1/2 | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of indication patient
PTF (peak to trough fluctuation ratio) | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of indication patient
CLss/F | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of indication patient
Vd,ss/F | 0 to 93 hr
  Liposome encapsulated amphotericin B and Unbound Amphotericin B of indication patient

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han S, Yim DS, Han S, Choi S, Cho SY, Lee R, Nho D, Baek HJ, Lee DG. Pharmacokinetic Equivalence of AmphosomTM, a Newly Developed Liposomal Amphotericin B, to AmbisomeⓇ. Clin Ther. 2026 Feb;48(2):186-195. doi: 10.1016/j.clinthera.2025.12.009. Epub 2026 Jan 8. PMID 41513548